CLINICAL TRIAL: NCT02557802
Title: Breadth of T-cell Responses After Heterologous Route Immunological Prime-boost Using Influenza Antigens as a Model System
Brief Title: T-cell Diversity Following Intranasal and Intramuscular Vaccines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CRC306C
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Nasal spray at day 0, intramuscular injection at day 28
  Interventions: Biological: Fluenz Tetra; Biological: Fluarix Tetra
- Group B (Experimental): Intramuscular injection at day 0, nasal spray at day 28
  Interventions: Biological: Fluenz Tetra; Biological: Fluarix Tetra

INTERVENTIONS:
Biological: Fluenz Tetra — Intranasal spray, 0.2 ml dose
Biological: Fluarix Tetra — Intramuscular injection, 0.5 ml dose

SUMMARY:
The investigators will explore in an experimental medicine healthy human model of immunisation, whether switching the route of sequential administration of licensed influenza vaccines can result in an immune response that is broader in its ability to recognise different substrains of influenza viruses. The investigators will do this by initially giving an immunisation with a nasal or an injected vaccine, and then switching subjects over to receive a second dose one month later (when the cellular component of immunity will have matured) via the opposite route (nasal->injected or injected->nasal). The investigators will use research assays that can map the different parts of the influenza virus that the vaccinated person's immune cells recognise at baseline, after the first immunisation, and then again after the second, to see if the breadth of the recognition has broadened to include new strains or virus components. Should this pilot study give an indication that the breadth has widened (rather than just a further boost to the same responses seen after the first immunisation) it will provide justification for a larger study in which statistical significance may be powered for observed changes.

The study is funded by ADITEC, which is a collaborative research programme that aims to accelerate the development of novel and powerful immunisation technologies for the next generation of human vaccines.

DETAILED DESCRIPTION:
This study is an Open-label, randomised, exploratory, hypothesis generating study.

Each participant will participate in the study for approximately two months. Recruitment aims to begin, on receipt of a favourable opinion from the ethics committee, in October/ November 2015, during the flu season.

There will be three outpatient visits during the study: Visit 1 will be screening and immunisation, Visit 2 will be immunisation, and Visit 3 will be an outpatient follow-up. All visits will take place at the Surrey Clinical Research Centre.

Written informed consent will be obtained after a participant is informed of the nature, significance, implications and risks of the study and prior to the commencement of any study specific procedures.

There will be two immunisations for each participant: one at Day 0 (visit 1) and the other at Day 28 (visit 2). After screening participants will be randomised to one of two treatment groups (n=15 in each group) and will receive a dose of the vaccine at the recommended dose level, according to the Summary of Product Characteristics, in the following orders:

Group A: Intranasal spray at day 0 followed by intramuscular injection at day 28

Group B: Intramuscular injection at day 0 followed by intranasal spray at day 28

Visit 1 (Day 0): At this visit informed consent will be obtained, demographic data and medical history recorded. Concomitant medications will be reviewed and a symptoms-directed physical examination will take place. Heart rate, blood pressure and oral temperature will also be recorded. A pregnancy test (urine) will be conducted where indicated. Participants will be assessed for inclusion and exclusion criteria. At this point if the participant is eligible they will be randomised to group A or B. Blood samples will be taken for serum and PBMC and they will be given the immunisation of either the nasal spray or the intramuscular injection depending on which group they are in.

Immunisation will be postponed if the person is suffering from an acute illness with an oral temperature ≥38.0°C on day of immunisation until the symptoms have resolved, and oral temperature is <38°C. Subsequent visits will be delayed by the same duration.

Visit 2 (Day 28): At visit two, medical history will be updated and there will be a review of concomitant medications. A symptoms-directed physical examination will also take place. Heart rate, blood pressure and oral temperature will also be recorded. A pregnancy test (urine) will be conducted where indicated. Participants will be again be assessed for inclusion and exclusion criteria. Blood samples will be taken for serum and PBMC and they will be given the immunisation of either the nasal spray or the intramuscular injection depending on which group they are in

Immunisation will be postponed if the person is suffering from an acute illness with an oral temperature ≥38.0°C on day of immunisation until the symptoms have resolved, and oral temperature is <38°C.

A visit window of -3 days or +7 days is acceptable for Visit 2 but should be avoided wherever possible and used only in a situation where a sample would otherwise be lost. Visit 3 should be rescheduled to maintain 28 days between visits.

Visit 3 (Day 56): At visit 3 there will be a review on concomitant medications and blood samples will be taken for serum and PBMC.

A visit window of -3 and +14 days is acceptable for Visit 3 but should be avoided wherever possible and used only in a situation where a sample would otherwise be lost. If participants cannot attend within this window then samples should be collected on the earliest date possible AFTER the expected visit window. These samples may be tested but will not be per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants aged 18-55 years inclusive at visit
2. Available for follow-up for the duration of the study.
3. If fertile female, willing to undergo urine pregnancy tests prior to immunisations.
4. Able to read and understand the Informed Consent Form (ICF), and understand study procedures and has signed the ICF.
5. Has not received any influenza vaccine in the 2015/16 influenza season.

Exclusion Criteria:

1. Any contraindication to receiving the study vaccines as detailed in the Summary of Product Characteristics.
2. Clinically significant medical condition that would interfere with study endpoints as determined by the study physician at screening.
3. Use of immunosuppressive/immunomodulating drugs orally or parenterally within 6 months of visit 1 or during the study follow-up period. Topical, inhaled and intranasal preparations are not excluded.
4. Currently participating in another clinical study with an investigational or non-investigational drug or device, or has participated in another clinical study within the 3 months preceding Visit 1.
5. Any condition that, in the investigator's opinion, compromises the participant's ability to meet protocol requirements or to complete the study.
6. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.
7. Positive pregnancy test on the day of immunisation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Breadth of T-cell responses | 8 months
  Breadth of T-cell responses to influenza antigens measured by increases in frequency and phenotype of T cells synthesising or secreting cytokines, or proliferating in response to in vitro stimulation with influenza antigens.

CONTACTS AND LOCATIONS:
Overall Officials: David Lewis, Principal Investigator — University of Surrey
Locations (1):
- Surrey Clinical Research Centre, Guildford, Surrey, United Kingdom